CLINICAL TRIAL: NCT04496622
Title: Comparison of Different Frequencies of Whole Body Vibration Training on Physical Function and Muscle Strength in Patients With Knee Osteoarthritis
Brief Title: WBV Training on Physical Function and Muscle Strength in Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00235 Anam Pervez
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Physical Function; Muscle Strength; Whole Body Vibration
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration Technique (Experimental): WBV training with the frequency of 16-25 Hz along with conventional treatment.
  Interventions: Other: WBV technique
- WBV Technique (Active Comparator): WBV training with the frequency of 26-35 Hz along with conventional treatment.
  Interventions: Other: Whole body vibration technique

INTERVENTIONS:
Other: WBV technique — Whole body vibration with frequency of 16-25 Hz were given from week 1-8 for 10 minutes/10 repetitions. Time were increased weekly Convention therapy were hot pack 10 minutes, stretching exercise (SLR) 10 repetition x 3 sets and quadriceps exercise 10 repetition x 3 sets.
  3 session/week for 8 weeks
  Arms: Whole Body Vibration Technique
Other: Whole body vibration technique — Whole body vibration with frequency of 26-35 Hz were given from week 1-8 for 10 minutes/10 repetitions. Time were increased weekly Convention therapy were hot pack 10 minutes, stretching exercise (SLR) 10 repetition x 3 sets and quadriceps exercise 10 repetition x 3 sets.
  3 session/week for 8 weeks
  Arms: WBV Technique

SUMMARY:
In this study compare different frequencies of whole body vibration training on physical function and muscle strength in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
This randomized controlled trial is to compare different frequencies of whole-body vibration (WBV) training on physical function and quadriceps muscle strength in patients with knee osteoarthritis and further will be researched which frequencies are effective for knee OA patients and how much WBV training is useful modality for knee osteoarthritic patients. This research will have significant effects in improving muscle strength and functional level of knee OA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Both genders
* Kellgren and Lawrance grade 2 and 3.
* Pain symptoms for at least 3 months
* Had no previous experience in WBV

Exclusion Criteria:

* Knee surgery in the past 6 months
* Patient with acute symptomatic knee OA
* Unable to walk unaided
* Diagnosed with other muscular and joint disease that affect the lower limb function
* Patient with any neurological conditions
* History of trauma to knee joint during last week.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 8 week
  Changes from base line WOMAC is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of hip and knee. It consists of 3 sections with the total score of 96
1 Repetition maximum (1 RM) | 8 week
  Changes from base line 1 RM measure muscle strength with maximum amount of weight that a person can possibly lift for one repetition

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 8 week
  Changes from baseline visual analog scale for pain starting from 0-10
Timed up and Go test (TUG) | 8 week
  Changes from baseline time up and go test to determine fall risk and measure the progress of balance, sit to stand and walking.
6 minute walk test | 8 week
  Changes from baseline 6 minute walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzuki Y, Iijima H, Tashiro Y, Kajiwara Y, Zeidan H, Shimoura K, Nishida Y, Bito T, Nakai K, Tatsumi M, Yoshimi S, Tsuboyama T, Aoyama T. Home exercise therapy to improve muscle strength and joint flexibility effectively treats pre-radiographic knee OA in community-dwelling elderly: a randomized controlled trial. Clin Rheumatol. 2019 Jan;38(1):133-141. doi: 10.1007/s10067-018-4263-3. Epub 2018 Aug 30. PMID 30167975
- [Background] Kus G, Yeldan I. Strengthening the quadriceps femoris muscle versus other knee training programs for the treatment of knee osteoarthritis. Rheumatol Int. 2019 Feb;39(2):203-218. doi: 10.1007/s00296-018-4199-6. Epub 2018 Nov 15. PMID 30430202
- [Background] Goh SL, Persson MSM, Stocks J, Hou Y, Welton NJ, Lin J, Hall MC, Doherty M, Zhang W. Relative Efficacy of Different Exercises for Pain, Function, Performance and Quality of Life in Knee and Hip Osteoarthritis: Systematic Review and Network Meta-Analysis. Sports Med. 2019 May;49(5):743-761. doi: 10.1007/s40279-019-01082-0. PMID 30830561
- [Background] Bacon KL, Segal NA, Oiestad BE, Lewis CE, Nevitt MC, Brown C, LaValley MP, McCulloch CE, Felson DT. Thresholds in the Relationship of Quadriceps Strength With Functional Limitations in Women With Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2019 Sep;71(9):1186-1193. doi: 10.1002/acr.23740. Epub 2019 Aug 6. PMID 30156759
- [Background] Roddy E, Zhang W, Doherty M, Arden NK, Barlow J, Birrell F, Carr A, Chakravarty K, Dickson J, Hay E, Hosie G, Hurley M, Jordan KM, McCarthy C, McMurdo M, Mockett S, O'Reilly S, Peat G, Pendleton A, Richards S. Evidence-based recommendations for the role of exercise in the management of osteoarthritis of the hip or knee--the MOVE consensus. Rheumatology (Oxford). 2005 Jan;44(1):67-73. doi: 10.1093/rheumatology/keh399. Epub 2004 Sep 7. PMID 15353613
- [Background] Park SY, Son WM, Kwon OS. Effects of whole body vibration training on body composition, skeletal muscle strength, and cardiovascular health. J Exerc Rehabil. 2015 Dec 31;11(6):289-95. doi: 10.12965/jer.150254. eCollection 2015 Dec. PMID 26730378
- [Background] Gerodimos V, Zafeiridis A, Karatrantou K, Vasilopoulou T, Chanou K, Pispirikou E. The acute effects of different whole-body vibration amplitudes and frequencies on flexibility and vertical jumping performance. J Sci Med Sport. 2010 Jul;13(4):438-43. doi: 10.1016/j.jsams.2009.09.001. Epub 2009 Oct 22. PMID 19853506
- [Background] Lai Z, Wang X, Lee S, Hou X, Wang L. Effects of whole body vibration exercise on neuromuscular function for individuals with knee osteoarthritis: study protocol for a randomized controlled trial. Trials. 2017 Sep 20;18(1):437. doi: 10.1186/s13063-017-2170-6. PMID 28931439